CLINICAL TRIAL: NCT04457271
Title: An EffectivenessTrial Examining a Novel Approach to Cognitive Remediation in Individuals With Post-Traumatic Stress Disorder (PTSD)
Brief Title: Goal Management Training in Individuals With PTSD
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Unfortunately, we have had to prioritize other studies and we do not have the resources required to carry out this study.
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); FDC Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 10037; 116096 (Registry Identifier: Western University's Research Ethics Board)
Record Dates: First submitted 2020-06-30; First posted 2020-07-07 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: PTSD; Post-traumatic Stress Disorder; Cognitive Impairment; Cognitive Dysfunction; Cognitive Deficit
Keywords: GMT; Goal Management Training; mindfulness; Cognitive Remediation
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Cognitive Dysfunction; Cognition Disorders

STUDY DESIGN:
Intervention Model Description: This study is an effectiveness trial investigating GMT as an intervention for both PTSD-related cognitive impairment/dysfunction, and PTSD symptoms themselves. Participants will be randomized to one of two conditions: GMT or wait list.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Goal Management Training (GMT) (Experimental): Participants in this arm will attend 9 weekly, 2-hour group GMT appointments.
  Interventions: Behavioral: Goal Management Training (GMT)
- Wait List (No Intervention): Participants in this arm will receive no treatment for approximately 21 weeks (at which point, they will be offered the same, standard GMT treatment).

INTERVENTIONS:
Behavioral: Goal Management Training (GMT) — GMT is a structured, short-term cognitive remediation program with an emphasis on mindfulness and practice in planning and completion of goal-oriented behaviours. The main objective of GMT is to help participants regain executive control in order to better define goals and monitor performance in achieving them. Sessions include instructional material, interactive tasks, discussion of patients' real-life deficits, and homework assignments. Mindfulness meditation is also incorporated for the purpose of developing the skill of bringing one's mind to the present to monitor ongoing behaviour, goal states, and the relationship between them, and for the development of attentional control. The program incorporates real-life examples to illustrate goal attainment failures and successes, as well as in-session practice of complex tasks that mimic real-life tasks - typically a challenge for individuals with executive function deficits (e.g., planning and set-shifting tasks).
  Arms: Goal Management Training (GMT)

SUMMARY:
This study will evaluate the effect of a manualized treatment (Goal Management Training, or GMT) on the cognitive impairments associated with PTSD (Post-Traumatic Stress Disorder), as well as any impact on PTSD symptems themselves. Participants will be randomized to either GMT group treatment, or a wait list condition.

DETAILED DESCRIPTION:
PTSD has an emotional impact on individuals, but it is also associated with impaired cognitive functioning (e.g., processing speed, attention, executive functioning). This study is an effectiveness trial investigating a cognitive remediation intervention (Goal Management Training, or GMT) that has been shown to improve the cognitive impairment observed in other populations (e.g., older adults). The present study will investigate the impact of GMT in adults experiencing PTSD (including frontline healthcare workers suffering from PTSD related to the COVID-19 pandemic) and its associated cognitive impairment. Participants will be randomly assigned to one of two treatment conditions - GMT, or a wait list condition (in which GMT will be postponed for approximately 21 weeks). Due to the pandemic, this study will be conducted primarily online (i.e., online assessments and treatment, with optional fMRI scans - functional magnetic resonance imaging). Once all assessments are complete, participants in the wait list condition will be able to begin GMT thelmselves.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of PTSD as determined by our baseline assessment
* Due to online nature: must have access to (and ability to use) a computer/tablet with a working microphone and camera (or webcam), reliable access to a secure internet connection, and access to a quiet, private space for the assessments and group sessions.
* Ability to provide informed consent
* Fluency in written and spoken English
* must be resident of Ontario (due to restrictions of professional licenses)

Exclusion Criteria for those opting in to fMRI scan:

* any implants, conditions, etc. that do not comply with 7T (Tesla) fMRI research safety standards (e.g., pacemaker, pregnancy/possible pregnancy)

Exclusion Criteria for study in general:

* history of significant head injury/lengthy loss of consciousness (e.g., a Glasgow Coma Scale Score < 15 at the time of incident as assessed retrospectively by participant)
* significant untreated medical illness
* history of neurological or neurodevelopmental disorder
* history of any pervasive developmental disorder
* any medical disorder known to adversely affect cognition within the last 12 months
* lifetime bipolar or psychotic disorder
* alcohol/substance abuse or dependence within the last 3 months
* extensive narcotic use (e.g., fentanyl, oxycodone, etc.), use of anti-cholinergics, anti-psychotics, psychostimulants, or benzodiazepines
* ECT (electroconvulsive therapy) within the last 12 months
* significant dissociative disorder (as determined by our baseline assessment)
* suicide attempt in last 6 months
* pregnancy (due to impact of hormones on cognitive abilities)
* hearing or vision issues that would interfere with effective online participation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-01 (Estimated); Primary Completion 2024-02 (Estimated); Study Completion 2024-02-01 (Estimated)

PRIMARY OUTCOMES:
Change in Sustained Attention to Response Task (SART) scores from baseline to post-treatment assessment | 9 weeks
  A computer-based go/no-go task that requires participants to withhold behavioral response to a single, infrequent target presented amidst a background of frequent non-targets. This task assesses inattentiveness, impulsivity, sustained attention, and vigilance.
Change in Sustained Attention to Response Task (SART) scores from post-treatment to 3-month follow-up assessment | 12 weeks
  A computer-based go/no-go task that requires participants to withhold behavioral response to a single, infrequent target presented amidst a background of frequent non-targets. This task assesses inattentiveness, impulsivity, sustained attention, and vigilance.
Change in score on Tower Test (part of Millisecond's online cognitive battery) from baseline to post-treatment assessment. | 9 weeks
  Assesses the participant's ability to act with forethought, and sequence behaviour in an orderly fashion to reach specific goals (i.e., executive functioning). Similar to the Tower of London test.
Change in score on Tower Test (part of Millisecond's online cognitive battery) from post-treatment to 3-month follow-up assessment. | 12 weeks
  Assesses the participant's ability to act with forethought, and sequence behaviour in an orderly fashion to reach specific goals (i.e., executive functioning). Similar to the Tower of London test.
Change in Difficulties in Emotion Regulation Scale (DERS) score from baseline to post-treatment assessment | 9 weeks
  A 36-item self-report measure that assesses difficulties with emotion regulation across six domains. A total score is derived by summing all the items - ranging from 36 to 180. Higher scores indicate greater dysfunction in emotion regulation.
Change in Difficulties in Emotion Regulation Scale (DERS) score from post-treatment to 3-month follow-up assessment | 12 weeks
  A 36-item self-report measure that assesses difficulties with emotion regulation across six domains. A total score is derived by summing all the items - ranging from 36 to 180. Higher scores indicate greater dysfunction in emotion regulation.
Change in Clinician Administered PTSD Scale (CAPS) score from baseline to post-treatment assessment | 9 weeks
  Gold standard, clinician administered PTSD assessment tool; min. score=0, max=80, with higher scores representing greater PTSD symptoms
Change in Clinician Administered PTSD Scale (CAPS) score from post-treatment to 3-month follow-up assessment | 12 weeks
  Gold standard, clinician administered PTSD assessment tool; min. score=0, max=80, with higher scores representing greater PTSD symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Ruth A. Lanius, MD, PhD, Principal Investigator — Lawson Research Institute
Locations (1):
- London Health Sciences Centre - University Hospital, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
Only coded data will be shared with co-investigators who are registered with the study's ethics board application.

REFERENCES:
- [Result] Boyd JE, Lanius RA, McKinnon MC. Mindfulness-based treatments for posttraumatic stress disorder: a review of the treatment literature and neurobiological evidence. J Psychiatry Neurosci. 2018 Jan;43(1):7-25. doi: 10.1503/jpn.170021. Epub 2017 Oct 2. PMID 29252162
- [Result] Meusel LA, Hall GB, Fougere P, McKinnon MC, MacQueen GM. Neural correlates of cognitive remediation in patients with mood disorders. Psychiatry Res. 2013 Nov 30;214(2):142-52. doi: 10.1016/j.pscychresns.2013.06.007. Epub 2013 Aug 30. PMID 23993991
- [Result] Lanius RA, Frewen PA, Tursich M, Jetly R, McKinnon MC. Restoring large-scale brain networks in PTSD and related disorders: a proposal for neuroscientifically-informed treatment interventions. Eur J Psychotraumatol. 2015 Mar 31;6:27313. doi: 10.3402/ejpt.v6.27313. eCollection 2015. PMID 25854674
- [Result] McKinnon MC, Boyd JE, Frewen PA, Lanius UF, Jetly R, Richardson JD, Lanius RA. A review of the relation between dissociation, memory, executive functioning and social cognition in military members and civilians with neuropsychiatric conditions. Neuropsychologia. 2016 Sep;90:210-34. doi: 10.1016/j.neuropsychologia.2016.07.017. Epub 2016 Jul 18. PMID 27444881